CLINICAL TRIAL: NCT00610662
Title: A Pilot Study: Measurement of Digital Colposcopy for Fluorescence Spectroscopy of Cervical Intraepithelial Neoplasia Using a Second Generation Device
Brief Title: Digital Colposcopy in Finding Cervical Intraepithelial Neoplasia in Patients With An Abnormal Pap Smear
Status: Withdrawn | Type: Observational
Why Stopped: Study modified and has been running as CDR0000581286 instead.
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000581295; BCCR-H07-01272 (Other: UBC-BCCA REB); P01CA082710 (NIH)
Record Dates: First submitted 2008-02-07; First posted 2008-02-08 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-04

CONDITIONS: Cervical Cancer; Precancerous Condition
Keywords: cervical cancer; cervical intraepithelial neoplasia grade 1; cervical intraepithelial neoplasia grade 2; cervical intraepithelial neoplasia grade 3
MeSH Terms: conditions — Uterine Cervical Neoplasms; Precancerous Conditions; Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
RATIONALE: Diagnostic procedures, such as digital colposcopy, may help doctors find and diagnose cervical intraepithelial neoplasia.

PURPOSE: This clinical trial is studying digital colposcopy to see how well it works in finding cervical intraepithelial neoplasia in patients with an abnormal Pap smear.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify potential improvements for a noninvasive method of diagnosing cervical dysplasia and neoplasia using the Multispectral Digital Colposcope (MDC), a device that uses fluorescence and reflectance spectroscopy to compare images with histopathologic mapping of the cervical epithelium.
* To measure MDC images in vivo of the cervix using a modified device that makes measurements in seconds rather than over 2 minutes before and after acetic acid.
* To evaluate, preliminarily, the effect of the fading of acetic acid in the image contrast obtained over time to see if this fading can predict the grade of intraepithelial neoplasia.
* To evaluate mapping of the cervix so that software can reconstruct the cervical epithelial map to compare the map with routine colposcopic images as well as with those from the MDC.
* To compare, preliminarily, MDC performance with colposcopy and pathologic analysis of tissue removed after colposcopy in the form of the loop electrosurgical excision procedure (LEEP).

OUTLINE: This is a multicenter study.

Patients undergo routine colposcopy as part of their regular colposcopic evaluation. The digital colposcope is used to take images of the vagina and cervix, pre- and post-acetic acid, using white, green, and blue light. Colposcopically abnormal areas are biopsied; a normal area may also be biopsied. Patients undergoing loop electrosurgical excision procedure (LEEP) may undergo one additional biopsy of a colposcopically normal site.

ELIGIBILITY:
Criteria

Inclusion criteria:

* Included subjects will be ≥18 years old.
* Included subjects will not be pregnant.
* Included subjects will have a negative urine pregnancy test.
* Included subjects will be scheduled for colposcopy and/or LEEP treatment at the VGH Women's Clinic.
* Included subjects will indicate understanding of the study.
* Included subjects will provide informed consent to participate.

Exclusion criteria:

* Individuals <18 years old will be excluded.
* Pregnant individuals will be excluded.
* Individuals that have had an operation to remove their cervix will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Identification of potential improvements for a noninvasive method of diagnosing cervical dysplasia and neoplasia using the Multispectral Digital Colposcope (MDC)
Measurement of MDC images in vivo of the cervix
Effect of the fading of acetic acid in the image contrast obtained over time and its prediction of the grade of intraepithelial neoplasia
Mapping of the cervix and comparison of map with routine colposcopic images as well as with those from the MDC
Comparison of MDC performance with colposcopy and pathologic analysis of tissue removed after colposcopy in the form of the loop electrosurgical excision procedure (LEEP)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas G Ehlen, M.D., Principal Investigator — British Columbia Cancer Agency, Vancouver General Hospital
Locations (1):
- BC Cancer Research Centre, Vancouver, British Columbia, Canada